## Statistical Analysis Plan Date: 12/21/2021

NCT04263987

## **Evaluation of the Moses Laser for Prostate Enucleation**

Nicholas Kavoussi, MD

Clinical Instructor of Urologic Surgery Vanderbilt University Medical Center Department of Urologic Surgery

## **Power and Statistical Analysis**

Power analysis was performed for sample size estimation based on prior reports from the literature, which previously estimated a 20% improvement in operative time when performing M-HoLEP. A sample size of 60 subjects had greater than 80% power to detect this change with  $\alpha$ =0.05. Continuous and categorical variables were compared using the Student T-test (2-tailed) and Fisher exact test, respectively. Multiple linear regression was performed to evaluate for the effect of the MOSES technique on operative time controlling for age, Charlson comorbidity index, change in hematocrit, and the amount of prostatic tissue enucleated. All testing was performed with p <0.05 as significant. All analyses were conducted in Stata 14.2 (StataCorp, College Station, Texas).